CLINICAL TRIAL: NCT04205617
Title: Living Hungry Healthy Foods Prescription Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Health Care District of Palm Beach County (Unknown); South Florida Hunger Coalition (Unknown); Jupiter Medical Center (Other); MyClinic, Inc (Unknown); FoundCare Inc. (Unknown); Living Hungry, Inc. (Unknown)
Responsible Party: Principal Investigator, Dariush Mozaffarian, Dean - Friedman School, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13491
Record Dates: First submitted 2019-12-16; First posted 2019-12-19 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus
Keywords: Produce prescription; Food insecurity; Nutrition education
MeSH Terms: conditions — Diabetes Mellitus | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Pre/post quasi experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Food Prescription (Experimental): Participants receive services through the Living Hungry program for food insecure diabetic patients.
  Interventions: Other: produce prescription and nutrition education

INTERVENTIONS:
Other: produce prescription and nutrition education — Participants will receive diabetic appropriate groceries, diabetes education classes led by volunteer doctors and nurses, cooking demonstrations, shared meals, 1:1 and group coaching by dietitians.
  Other Names: medically tailored food

SUMMARY:
This study is a pre/post, pilot evaluation of the 4-month, Living Hungry program for food-insecure patients with uncontrolled diabetes. The program provides free produce, whole grains and legumes to participants and their household every-other week, in addition, to nutrition education and glucose monitoring devices. The study is analyzing diabetes management indicators, including HbA1c, dietary quality, food insecurity, and medication adherence, plus health care utilization.

DETAILED DESCRIPTION:
The Living Hungry Collaborative, in partnership with the South Florida Hunger Coalition, previously operated a pilot program, Fresh Food Farmacy, staged from June 1, 2018, to September 29, 2018. The program consisted of nine Eat Well Pop-Up Pantry events at the My Clinic in Jupiter, Florida, serving 104 patients and feeding approximately 300 people including their families. Each set of groceries contained two weeks' worth of "medically tailored" groceries for diabetic-friendly meals for food-insecure patients diagnosed with diabetes or prediabetes. All clients involved in the intervention were referred by staff at the same four clinics that will participate in this study: My Clinic, C.L. Brumback Clinic in Jupiter, Jupiter Medical Center, and FoundCare. The Living Hungry Collaborative has an ongoing program to further evolve and test the "Fresh Food Farmacy", renamed as the Healthy Food Prescription Program intervention in Palm Beach County, for food-insecure, diabetic patients.

In addition to receiving diabetic appropriate groceries at the former Fresh Food Farmacy events, clients will be engaged in diabetes education classes led by volunteer doctors and nurses, cooking demonstrations, shared meals, 1:1 and group coaching by nutritionists and dietitians on best choices from a menu for diabetics, and tasting new recipes with produce from the pop-up event. The pilot program allowed Living Hungry to fine-tune the patient referral process, distribution logistics, and establish strong partnerships required for the next phase of the program. However, gaps exist to understand the extent to which the program design is improving the health of the participating diabetic patients.

Living Hungry will partner with Tufts University to conduct an evaluation of this existing program on key health outcomes that concern the partner clinics, specifically: biomarkers including Hemoglobin A1C, BMI, blood pressure, lipid profile, health care utilization including medication use, hospitalizations, emergency department visits, and health care costs, plus dietary quality, food insecurity, medication use, and quality of life indicators. The study is a pilot evaluation, implementing a quasi-experimental, pre/post study design.

The Living Hungry Healthy Foods Prescription Program is a community-based program that will be available to individuals whether or not they participate in the evaluation by Tufts University. This program is using the same referral and data collections procedures as the pilot, which include having physicians at the partner clinics refer patients with HbA1C levels greater than 8.0 mmol/mol and who are food insecure to Living Hungry to participate in the program. In addition, Living Hungry will again collect data on HbA1c, BMI, blood pressure, lipid profiles, and distribute a survey to participants.

ELIGIBILITY:
Inclusion Criteria:

1. Referred patient from one of four medical partners: My Clinic, C.L. Brumback Clinic, FoundCare and Jupiter Medical Center and has been a patient for at least one-year.
2. Diabetic with A1C over 8.0
3. Adults 18 years of age or older
4. Food-insecure

Exclusion Criteria:

1. Referred patients with HbA1c levels below 8.0 mmol/mol
2. Minors
3. Adults with severe mental illness who cannot provide informed consent, unless they have present a lawful caregiver or power of attorney.
4. Anyone who does not plan on staying in West Palm Beach for the next 4 months.
5. Pregnant women (can still receive services through the program but will not be included in the analysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | pre/post change in HbA1c in participants from baseline to completion of the program at 4 months
  will be measured by blood draws at first and last program event

SECONDARY OUTCOMES:
Change in frequency of hospitalizations | pre/post change in hospitalizations in participants from baseline to one month after completion of the program
  will be measured through surveys and data from electronic medical records
Change in frequency of emergency department admissions | pre/post change in emergency department admissions in participants from baseline to one month after completion of the program
  will be measured through surveys and data from electronic medical records
Change in total health care costs | pre/post change in total health care costs in participants from baseline to one month after completion of the program
  will be measured through data from hospital records
Change in food insecurity | pre/post change in food insecurity in participants from baseline to completion of the program at 4 months
  Food insecurity will be measured using the USDA 9-question food insecurity screener
Change in daily servings of fruits and vegetables | pre/post change in daily servings of fruits and vegetables in participants from baseline to completion of the program at 4 months
  Will be assessed through a food frequency questionnaire modeled off the USDA FINI assessment tool
Change in daily servings of whole grains | pre/post change in daily servings of whole grains in participants from baseline to completion of the program at 4 months
  Will be assessed through a food frequency questionnaire modeled off the USDA FINI assessment tool
Change in daily servings of lean proteins | pre/post change in daily servings of lean proteins in participants from baseline to completion of the program at 4 months
  Will be assessed through a food frequency questionnaire modeled off the USDA FINI assessment tool and includes: nuts, seeds, legumes, poultry, and fish.
Change in daily servings of sugary snacks and drinks | pre/post change in daily servings of sugary snacks and drinks in participants from baseline to completion of the program at 4 months
  Will be assessed through a food frequency questionnaire modeled off the USDA FINI assessment tool and includes: sugar sweetened beverages, pastries, cookies, cakes, candy, and other sweets
Change in medication adherence | pre/post change in medication adherence in participants from baseline to completion of the program at 4 months
  Measured as a composite score that will be assessed through a survey. Components include: frequency of sacrificing medication purchases for other household needs (such as food, utilities) and change in medication use.
Change in adhering to recommended diabetes management plan | pre/post change in in adhering to recommended diabetes management in participants from baseline to completion of the program at 4 months
  Measured as a composite scale that will be assessed through a survey. Components include frequency in which participants followed the recommendations of their physicians to manage their diabetes.
Change in blood LDL level | pre/post change in systolic blood LDL levels in participants from baseline to completion of the program at 4 months
  measured at first and last program event through a blood draw
Change in systolic blood pressure | pre/post change in systolic blood pressure in participants from baseline to completion of the program at 4 months
  measured at first and last program event
Change in diastolic blood pressure | pre/post change in diastolic blood pressure in participants from baseline to completion of the program at 4 months
  measured at first and last program event

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Mozaffarian, MD, DrPH, Principal Investigator — Tufts University Friedman School of Nutrition Science and Policy
Locations (1):
- Living Hungry, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No